CLINICAL TRIAL: NCT01743183
Title: Influence of Respiratory Muscle Training in Elderly Hypertensive Women With Respiratory Muscle Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Foundation for research support from the state of Rio Grande do Norte (FAPERN) (Unknown)
Responsible Party: Principal Investigator, Patra-cia Angelica de Miranda Silva Nogueira, Patrícia Angélica de Miranda Silva Nogueira, Universidade Federal do Rio Grande do Norte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05135912.8.0000.5537
Record Dates: First submitted 2012-11-12; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension | interventions — Speech Reception Threshold Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- threshold (Experimental): Held inspiratory muscle strengthening for 5 weeks with Threshold, charging 30% of maximal inspiratory pressure, 7 days a week, one supervised and unsupervised 6.
  Interventions: Device: Threshold

INTERVENTIONS:
Device: Threshold — The load adjustment was done weekly by a single examiner.

SUMMARY:
This study aims to evaluate pulmonary function and respiratory muscle strength in a group of elderly women with hypertension before and after a respiratory muscle training.

DETAILED DESCRIPTION:
It is a respiratory muscle training using the Threshold for 5 weeks, with a load of 30% of maximal inspiratory pressure obtained in manometer for 30 minutes daily. Furthermore, the assessment includes: test 6-minute walk, the quality of life questionnaire, MINICHAL, the IPAQ short version, manometer and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hypertension controlled by antihypertensive;
* aged between 60 and 80 years;
* absence of dementia or cognitive impairments that limit tests;
* absence of recent myocardial infarction;
* absence of musculoskeletal limitations that limit tests;
* availability of time on training days.

Exclusion Criteria:

* clinical instability;
* inability to perform any test.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
manovacuometry | 6 weeks
  Evaluates indirectly respiratory muscle strength.

SECONDARY OUTCOMES:
spirometry
  Assesses lung function

OTHER OUTCOMES:
quality of life
  Assesses the influence of hypertension on the quality of life of target
functional capacity
  assesses the cardiopulmonary capacity at sub-maximal
IPAQ
  assesses the level of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Nogueira, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil